CLINICAL TRIAL: NCT05265949
Title: The Effects of Dietary and Physical Activity Interventions on Tinnitus Symptoms: An RCT
Brief Title: The Effects of Weight Loss on Tinnitus Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, ümüş özbey yücel, Clinical Researcher of the Ankara University Audiology Department, Ankara University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraUniv
Record Dates: First submitted 2021-12-13; First posted 2022-03-04 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Subjective Tinnitus; Obesity
Keywords: tinnitus; diet; physical activity
MeSH Terms: conditions — Tinnitus; Obesity; Motor Activity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- diet+physical activity (Experimental): diet+physical activity
  Interventions: Behavioral: diet and physical activity intervention
- diet (Experimental): diet
  Interventions: Behavioral: diet and physical activity intervention
- physical activity (Experimental): physical activity
  Interventions: Behavioral: diet and physical activity intervention
- control (No Intervention): control

INTERVENTIONS:
Behavioral: diet and physical activity intervention — Dietary intervention: Preparation and follow-up of diet program Physical activity intervention: Step count monitoring
  Arms: diet; diet+physical activity; physical activity

SUMMARY:
Subjective tinnitus is the perception of irregular sound at different frequencies. Although the underlying cause of tinnitus is unclear, increased body weight is known to increase tinnitus symptoms. This study aimed to determine the effects of dietary and physical activity interventions on tinnitus symptoms. Sixty-three obese subjects with tinnitus aged 20 to 65 years were divided into diet + physical 8 activity (P.A.), diet, P.A., and control groups. Dietary and anthropometric records, Tinnitus Handicap 9Inventory (THI), Beck Depression Inventory (BDI), Short-Form Health Survey (SF-36), and Visual Analogue Scale (VAS) of all individuals were compared at the baseline and at the end of the study.

DETAILED DESCRIPTION:
Although the underlying cause of tinnitus is unclear, increased body weight is known to increase tinnitus symptoms. The present study aimed to determine the effects of dietary and physical activity interventions on tinnitus symptoms.

Sixty-three obese subjects with tinnitus aged 20 to 65 years were divided into diet + physical activity (P.A.) (n = 15), diet (n = 16), P.A. (n = 15), and control (n = 17) groups. Dietary records, anthropometric measurements, Tinnitus Handicap Inventory (THI), Beck Depression Inventory (BDI), Short-Form Health Survey (SF-36), and Visual Analogue Scale (VAS) of all individuals were recorded and compared at the baseline and at study completion.

ELIGIBILITY:
Inclusion Criteria:

* obese

Exclusion Criteria:

* diagnosed with tinnitus

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Weight Loss | At the end of the 3 months
  BMI (kilogram/ metre2 (kg/m2))
Tinnitus Severity | At the end of the 3 months
  Desibel (dB)
Tinnitus Frequency | At the end of the 3 months
  Heartz (hz)

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Score | At the end of the 3 months
  The score ranges from 1 to 10 points, with increasing score reflecting more discomfort
Quality of Life Score | At the end of the 3 months
  The score ranges from 0 to 100 points, with an increased score reflecting improved quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Ümüş Özbey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No